CLINICAL TRIAL: NCT05116020
Title: Swiss Chiropractic Cohort (Swiss ChiCo) Study: Prospective Clinical Cohort of Patients With Musculoskeletal Pain
Brief Title: Swiss Chiropractic Cohort (Swiss ChiCo) Study: Patient Cohort
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other); University of Southern Denmark, Department of Sports Science and Clinical Biomechanics (Unknown); Swiss Chiropractic Association (ChiroSuisse) (Unknown); Swiss Chiropractic Patient Association (Pro Chiropractic Switzerland) (Unknown)
Responsible Party: Sponsor
Other Study IDs: SwissChiCo-Patient
Record Dates: First submitted 2021-09-08; First posted 2021-11-10 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Musculoskeletal Pain
Keywords: Chiropractic; Musculoskeletal health; Musculoskeletal pain; Health care quality
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chiropractic patient participants: Usual chiropractic care
  Interventions: Other: Usual chiropractic care

INTERVENTIONS:
Other: Usual chiropractic care — Usual chiropractic care in Switzerland can include spinal manual therapy, soft-tissue therapy, use of electric therapeutic modalities (low level laser therapy, therapeutic ultrasound, interferential current), acupuncture, prescription medication, exercise, education and reassurance.

SUMMARY:
The Swiss chiropractic patient cohort (Swiss ChiCo) study is a nationwide research project which aims to describe the characteristics of patients presenting to Swiss chiropractors, assess the clinical course of patients with musculoskeletal pain, and examine the feasibility for performing a larger subsequent cohort study.

DETAILED DESCRIPTION:
The chiropractic scope of practice within Switzerland includes the diagnosis and management of musculoskeletal (MSK) pain conditions through manual medicine, prescription medication, and diagnostic imaging (radiography, ultrasound, CT, MRI). Common patient complaints presenting to Swiss chiropractic offices mirror this scope of practice, with low back pain and pelvic related pain being the most prevalent. This combination of clinical expertise and access to a MSK pain patient population allows chiropractic health care centres to become useful "real-world" primary care settings to further understand the current management and clinical course of MSK pain conditions in Switzerland, and to identify practice gaps and opportunities for Swiss MSK primary health care quality improvement.

This study aims to describe the characteristics of patients with new conservative healthcare seeking for MSK pain presenting to Swiss chiropractors, assess the clinical course of these patients over 12 weeks, and examine the feasibility for performing a larger subsequent prospective electronic cohort study using the newly established Swiss ChiCo practice-based research network (PBRN) and clinical cohort methodological framework.

Participating chiropractors will recruit consecutive patients from community-based chiropractic practices into a 12-week observational prospective electronic cohort study. Patient participants will be asked to complete 5 electronic surveys over 12-weeks. The first survey will be provided to patient participants prior to their initial chiropractic assessment. Subsequent questionnaires will be provided 1-hour, 2-weeks, 6-weeks, and 12-weeks after the initial visit. This patient cohort study represents a collaborative effort of international researchers, Swiss chiropractic clinicians, and the chiropractic patient and clinical associations in Switzerland (Pro Chiropractic Switzerland and ChiroSuisse). The survey design and study implementation procedures have been conceptualized through stakeholder consultation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Seeking new conservative health care for a musculoskeletal pain condition at a Swiss chiropractic clinic (ie, not having received participant-reported chiropractic care, physiotherapy, osteopathy, or massage therapy for the musculoskeletal complaint in the past 1 month and not a follow-up visit)
* Consent to chiropractic treatment
* Proficient in German, French, Italian, or English
* Active email account
* Willing to complete electronic study questionnaires

Exclusion Criteria:

* Presenting with red-flag symptoms (i.e., saddle anesthesia, loss of bowel and/or bladder control, history of major trauma, fracture, fever, severe or rapidly progressive neurologic deficit, sudden unexpected weight loss)
* Presenting with non-musculoskeletal pain condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons presenting to chiropractic clinic seeking new conservative health care for a musculoskeletal pain condition in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in musculoskeletal pain impact | Baseline; 1-hour after initial visit; 2-, 6-, 12-weeks
  Assessment via Pain, Enjoyment, and General Activity scale (PEG scale, 0-10). A higher score reflects worse outcome (worse pain intensity and interference)
Change in musculoskeletal health status | Baseline; 1-hour after initial visit; 2-, 6-, 12-weeks
  Assessment via musculoskeletal health questionnaire (MSK-HQ, 0-56). A higher score reflects better musculoskeletal health status
Invited patient participation proportion | Baseline
  Proportion of invited patients who agree to participate (feasibility outcome)
Change in participant follow-up and retention | Baseline; 1-hour after initial visit; 2-, 6-, 12-weeks
  Proportion of enrolled participants who complete follow-up surveys (feasibility outcome)

SECONDARY OUTCOMES:
Reasons for non-participation | Baseline
  Reasons for invited participant non-participation (no email address, unfamiliar with electronic or internet tools, lack of time, lack of interest in the study, data privacy concerns, other)
Factors associated with non-response | Baseline and 12-weeks
  A multivariable logistic regression analysis will be performed to assess the association between the participant factors (listed below) and non-response (versus response) at 12-weeks follow-up. Participant factors that will be assessed are: age (reported in years), sex (reported as male and female), medication use for MSK pain (reported as prescription medication, non-prescription medication, and no medication use), current MSK pain condition episode duration (dichotomised as acute [< 3 months duration] and chronic [≥ 3 months duration]), MSK pain impact (PEG scale, 0-10), and MSK health status (MSK-HQ, 0-56) collected at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Hincapié, DC PhD, Principal Investigator — Balgrist University Hospital and University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data may be made available for research purposes. Requests, including a synopsis of the study plan, can be addressed to the central contact person.

REFERENCES:
- [Background] Lalji R, Hofstetter L, Kongsted A, von Wyl V, Puhan MA, Hincapie CA. Swiss chiropractic practice-based research network and musculoskeletal pain cohort pilot study: protocol of a nationwide resource to advance musculoskeletal health services research. BMJ Open. 2022 Jul 13;12(7):e059380. doi: 10.1136/bmjopen-2021-059380. PMID 35831057
- [Background] Lalji R, Hofstetter L, Kongsted A, von Wyl V, Puhan MA, Hincapie CA. The Swiss chiropractic practice-based research network: a population-based cross-sectional study to inform future musculoskeletal research. Sci Rep. 2023 Apr 6;13(1):5655. doi: 10.1038/s41598-023-32437-3. PMID 37024506
- [Derived] Lalji R, Hofstetter L, Kongsted A, von Wyl V, Braun J, Puhan MA, Hincapie CA; Swiss ChiCo Clinicians Group. Swiss chiropractic cohort (Swiss ChiCo) pilot study: feasibility for a musculoskeletal cohort study conducted within a nationwide practice-based research network. Eur Spine J. 2024 May;33(5):2068-2078. doi: 10.1007/s00586-024-08175-z. Epub 2024 Mar 13. PMID 38480624
- See also: Musculoskeletal Epidemiology Research Group, Balgrist University Hospital, Project webpage — https://www.balgrist.ch/en/research/research-units/research-orthopaedics/musculoskeletal-epidemiology-research/research-projects/